CLINICAL TRIAL: NCT07253298
Title: Effects of Kegel Exercise Combined With a Single Biofeedback Intervention on Bowel Function, Emotional Distress, and Quality of Life in Patients After Rectal Cancer Surgery
Brief Title: The Effects of Kegel Exercise Combined With Biofeedback Therapy on Bowel Function Recovery, Emotional Distress, and Quality of Life in Patients Following Low Anterior Resection for Rectal Cancer
Acronym: BFT in LARS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202502004RINB
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Rectal Cancer; Low Anterior Resection Syndrome; LARS - Low Anterior Resection Syndrome
Keywords: Kegel exercise; Biofeedback therapy; Bowel dysfunction; Emotional distress; Quality of life; Rectal cancer patients; Pelvic floor muscle training; Rehabilitation
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome; Intestinal Diseases | interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: This study uses a two-arm parallel group design comparing Kegel exercise combined with a single biofeedback therapy versus Kegel exercise alone.
Who Masked: Outcomes Assessor
Masking Description: Description: Data collectors were blinded to participant group assignment to reduce potential information bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kegel Exercise with Biofeedback Therapy (Experimental)
  Interventions: Behavioral: Kegel Exercise with Biofeedback
- Kegel Exercise Only (Active Comparator)
  Interventions: Behavioral: Kegel Exercise Only

INTERVENTIONS:
Behavioral: Kegel Exercise with Biofeedback — A single 30-minute non-invasive EMG biofeedback session will guide participants to correctly contract and relax pelvic floor muscles using real-time visual and auditory feedback. Conducted by trained healthcare staff in the physical therapy center, with additional outpatient or ward instruction if needed. After the session, participants perform home-based Kegel exercises for 8 weeks (3-5 times/day, 6-8 contractions/set, hold 5-10 sec, relax 10 sec, ≥5 days/week). Research staff will follow up every 1-2 weeks by phone to monitor adherence and adjust intensity. If stable 5-sec contractions are achieved, duration or frequency may increase; if fatigue, abdominal pressure, or discomfort occurs, training will be reduced or paused for safety.
  Other Names: Kegel Exercise with Biofeedback (Kegel + BFT)
  Arms: Kegel Exercise with Biofeedback Therapy
Behavioral: Kegel Exercise Only — Participants in the control group will receive a single 30-minute session of verbal instruction and demonstration on Kegel exercise by trained medical personnel, without the use of any biofeedback device. The provider, setting, duration, exercise dosage, and follow-up schedule are identical to those in the experimental group.
  Other Names: Kegel Exercise
  Arms: Kegel Exercise Only

SUMMARY:
This randomized controlled trial aims to evaluate the effects of combining Kegel exercise with a single biofeedback session on bowel function, emotional distress, and quality of life in patients who have undergone low anterior resection (LAR) for rectal cancer. Low anterior resection syndrome (LARS) is a common postoperative complication following LAR, characterized by increased stool frequency, urgency, and incontinence, which can significantly impair patients' psychological well-being and daily quality of life. Participants will be randomly assigned to one of two groups: (1) Kegel exercise combined with one non-invasive biofeedback session, or (2) Kegel exercise alone. Both groups will perform home-based Kegel exercises for eight weeks. The study aims to determine whether the combined biofeedback and Kegel exercise intervention results in greater improvements in bowel control, emotional well-being, and quality of life compared with Kegel exercise alone.

DETAILED DESCRIPTION:
Background:

Patients who undergo low anterior resection (LAR) for rectal cancer often experience low anterior resection syndrome (LARS), characterized by frequent bowel movements, urgency, and incontinence. These symptoms can cause considerable psychological distress and impair daily functioning. Pelvic floor muscle training (PFMT, commonly known as Kegel exercise) is a widely used bowel rehabilitation method; however, its effectiveness depends on patients' ability to perform the exercises correctly. Biofeedback therapy (BFT) provides real-time visual and auditory feedback to help patients better control pelvic floor muscle contractions and relaxations, thereby improving training precision.

Objective:

To examine whether combining a single biofeedback intervention with Kegel exercise produces greater improvements in bowel function, emotional distress, and quality of life than Kegel exercise alone in patients after low anterior resection for rectal cancer.

Methods:

This is a prospective randomized controlled trial (IRB No. 202502004RINB) to be conducted at National Taiwan University Hospital. A total of 66 eligible participants who have completed at least four weeks after LAR will be recruited. Participants will be randomized (1:1) into experimental and control groups using block randomization with block sizes of 4, 6, or 8.

The experimental group will receive one 30-minute session of non-invasive electromyographic biofeedback training to correct pelvic floor muscle contraction and relaxation techniques, followed by Kegel exercise instruction. The control group will receive only verbal instruction and demonstration of Kegel exercises without the use of biofeedback devices.

Both groups will continue home-based Kegel exercises for eight weeks, with a total follow-up period of twelve weeks. Assessments will be conducted at four time points: baseline (T0), 4 weeks (T1), 8 weeks (T2), and 12 weeks (T3).

Outcome Measures:

Primary outcome: Low Anterior Resection Syndrome Score (LARS Score). Secondary outcomes: Hospital Anxiety and Depression Scale (HADS), The World Health Organization Quality of Life Assessment-BREF Taiwan version (WHOQOL-BREF Taiwan version).

Expected Results:

The experimental group (Kegel exercise combined with single-session biofeedback) is expected to demonstrate greater improvements in bowel function, reduced emotional distress, and enhanced quality of life compared with the Kegel-only group.

Significance:

This study aims to establish a low-cost, non-invasive, and feasible postoperative rehabilitation approach to enhance bowel recovery and improve the quality of life in patients after rectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone their first low anterior resection (LAR) for rectal cancer, or LAR with temporary stoma reversal at least 4 weeks prior to enrollment.
* Age ≥ 18 years.
* Hemodynamically stable with stable vital signs.
* Conscious, able to communicate in Mandarin or Taiwanese, and capable of following verbal instructions to perform exercises.

Exclusion Criteria:

* Presence of a current intestinal stoma.
* Implanted cardiac pacemaker.
* Scheduled to receive postoperative adjuvant radiotherapy.
* History of psychiatric disorders (e.g., depression).
* Postoperative complications such as anastomotic leakage, intra-abdominal infection, or fistula formation.
* Unable to cooperate with or complete biofeedback training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Bowel Function Measured by the Low Anterior Resection Syndrome (LARS) Score | Baseline, 4 weeks, 8 weeks, and 12 weeks after intervention
  Bowel function will be assessed using the validated Low Anterior Resection Syndrome (LARS) score, which consists of five items evaluating incontinence, frequency, clustering, and urgency. The total score ranges from 0 to 42, with higher scores indicating more severe bowel dysfunction.

SECONDARY OUTCOMES:
Change in Emotional Distress Measured by the Hospital Anxiety and Depression Scale (HADS) | Baseline, 4 weeks, 8 weeks, and 12 weeks after intervention
  Emotional distress will be measured using the Hospital Anxiety and Depression Scale (HADS), which includes 14 items divided into two subscales: anxiety (HADS-A) and depression (HADS-D). Each subscale has a score range of 0-21, with higher scores indicating greater emotional distress.
The World Health Organization Quality of Life Assessment-BREF (WHOQOL-BREF) | Baseline, 4 weeks, 8 weeks, and 12 weeks after intervention
  Quality of life will be assessed using the WHOQOL-BREF Taiwan version, a 28-item instrument developed by the WHOQOL Group and culturally adapted for use in Taiwan. The scale measures four major domains-Physical Health, Psychological Health, Social Relationships, and Environment-as well as two national items relevant to local culture. Scores in each domain are transformed to a 4-20 scale, with higher scores indicating better perceived quality of life.

IPD SHARING:
Plan to Share IPD: No